CLINICAL TRIAL: NCT01950689
Title: A Randomised Placebo-controlled Trial of Synchronous NIMorazole Versus RADiotherapy Alone in Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma Not Suitable for Synchronous Chemotherapy or Cetuximab)
Brief Title: NIMRAD (A Randomised Placebo-controlled Trial of Synchronous NIMorazole Versus RADiotherapy Alone in Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma Not Suitable for Synchronous Chemotherapy or Cetuximab)
Acronym: NIMRAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Yamina Ainaoui, Clinical Trials Manager, The Christie NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFTSp032, 11_DOG08_53
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Nimorazole; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo given in parallel with radiotherapy for 6 weeks.
  Interventions: Radiation: Radiotherapy
- Nimorazole (Experimental): Nimorazole given in parallel with radiotherapy for 6 weeks
  Interventions: Drug: Nimorazole; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Nimorazole
  Arms: Nimorazole
Radiation: Radiotherapy

SUMMARY:
The purpose of this study is to see whether adding Nimorazole to standard radiotherapy benefits patients with locally advanced head and neck squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed (newly diagnosed/ not recurrent) head and neck squamous cell carcinoma; all primary subsites EXCEPT nasal cavity, oral cavity, nasopharynx and paranasal sinus (i.e. oropharynx, hypopharynx, larynx are allowed)
* Stage T3/T4 N0; any node +ve case including T1 node +ve; T2N0 base of tongue/hypopharynx
* Patients suitable for definitive radiotherapy. Block dissections may be performed pre-RT for N2/N3 disease
* WHO status 0-2
* Patient fit and able to undergo RT with nimorazole and be expected to complete treatment
* Absence of another disease or previous malignancy which is likely to interfere with the treatment or assessment of response
* No evidence of distant metastases (M0)
* Unable to tolerate/unlikely to benefit from platinum chemotherapy or monoclonal antibody therapy
* Women must be postmenopausal (no menstrual period for a minimum of 1 year) or have a negative serum pregnancy test on entry in the study (even if surgically sterilised) and be using an adequate contraception method. This must be continued for 1 week after completion of nimorazole, unless child bearing potential has been terminated by surgery/radical radiotherapy
* Men must be willing to use an adequate method of contraception during treatment and until 1 week after nimorazole
* Greater than 18 years of age; no upper age limit
* Available for follow up within the United Kingdom
* Adequate renal and liver function - absolute neutrophil count >=1.5 x 109/L, creatinine <=2x ULN, platelets > 100x109/L, total bilirubin <=2 x ULN, AST or ALT <3 x ULN
* The capacity to understand the patient information sheet and the ability to provide written informed consent
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures

Exclusion Criteria:

* Patients with T1N0 tumours or those within the nasopharynx, nasal cavity or sinus, oral cavity; T2No larynx and tonsil; unknown primary cancer.
* Any prior chemotherapy in the last 6 months or RT within the planned radiation field
* Presence of any life threatening illness such as unstable angina or severe chronic obstructive pulmonary disease
* Mental disability or patient otherwise unable to give informed consent and/or complete patient questionnaires
* Hb <100 g/l (patients with anaemia may be transfused to bring Hb levels to >100 g/l within 1 week of treatment start. Please repeat Hb following transfusion to confirm now eligible)
* Peripheral neurophathy as assessed clinically (CTCAE >=2)
* Use of any investigational drug within 30 days prior to screening
* Severe and/or uncontrolled medical disease
* Any malabsorption syndrome (i.e. partial gastrectomy, small bowel resection, Crohn's disease or ulcerative colitis)
* Use of Lithium or Phenobarbitone during the study
* Patients who are breastfeeding or pregnant
* Previous malignancy within 5 years (except BCC, in-situ Ca e.g. of the cervix)
* Previous definitive surgery to primary site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2014-09-11 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
Locoregional Control in patients with more hypoxic tumours (the enriched population) | 12 weeks post treatment
  To examine whether patients with locally advanced head and neck squamous cell carcinoma unsuitable for either cisplatin chemotherapy or monoclonal antibody therapy benefit from the addition of nimorazole to standard definitive radiotherapy in terms of increased locoregional control without additional serious toxicity.

SECONDARY OUTCOMES:
Overall survival (enriched sub-group) | Date of death for patient, month 60.
Cancer-specific survival (enriched sub-group) | follow up month 60
Disease-free survival (enriched sub-group) | follow up month 60
Cumulative incidence of loco-regional failure | follow up month 60
Acute toxicity (all patients) | baseline, week 1, 2, 3, 4, 5, 6, follow up month 1.5 and 3
Hypoxia signature prediction of nimorazole benefit (all patients) | screening
Quality of life (enriched sub-group) | baseline, week 6, month 6, 12, 18, 24, 36 of follow up
Late toxicity (all patients) | baseline, follow up month 6, 12, 18, 24, 36

CONTACTS AND LOCATIONS:
Overall Officials: David Thomson, Principal Investigator — The Christie NHS Foundation Trust
Locations (21):
- United Kingdom (21):
  - Cheltenham General Hospital, Cheltenham, Gloucestershire
  - Clatterbridge Centre for Oncology, Bebington, Merseyside
  - St James' Hospital, Leeds, West Yorkshire
  - Belfast City Hospital, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - Bristol Haematology and Oncology centre, Bristol
  - Addenbrookes Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - University Hospitals Coventry and Warwickshire, Coventry
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - The Royal Surrey County Hospital, Guildford
  - Leicester Royal Infirmary, Leicester
  - University College London Hospital, London
  - The Royal Marsden, London
  - The Christie NHS Foundation Trust, Manchester
  - The James Cook University Hospital, Middlesbrough
  - Nottingham University Hospitals, Nottingham
  - Weston Park Hospital, Sheffield
  - Singleton Hospital, Swansea
  - York Hospital, York